CLINICAL TRIAL: NCT07385664
Title: A Phase II Study of Neoadjuvant Chemoimmunotherapy or Concurrent Chemoradiotherapy Guided by Post-Chemoimmunotherapy FAPI-PET/CT
Brief Title: Neoadjuvant Chemoimmunotherapy or Chemoradiotherapy in ESCC
Acronym: FAIR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ji Yongling (Other)
Responsible Party: Sponsor-Investigator, Ji Yongling, Clinical Professor, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2025-424
Record Dates: First submitted 2025-05-20; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Resectable Esophageal Cancer
Keywords: FAPI-PET/CT; Resectable Esophageal Cancer; Neoadjuvant Therapy
MeSH Terms: interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy + PD-1 inhibitor (Experimental): Patients initially received two cycles of neoadjuvant chemotherapy in combination with immunotherapy. The chemotherapy protocol consisted of albumin-bound paclitaxel (260mg/m2, with a maximum dose of 400mg) + carboplatin (AUC=5). Sintilimab was employed for immunotherapy at a fixed dose of 200mg.
  Interventions: Combination Product: Neoadjuvant Chemoimmunotherapy or Concurrent Chemoradiotherapy

INTERVENTIONS:
Combination Product: Neoadjuvant Chemoimmunotherapy or Concurrent Chemoradiotherapy — FAPI-PET/CT was carried out between days 15 and 22 after two cycles of chemoimmunotherapy. If the FAPI-PET/CT results indicated that the SUVmax of the primary lesion decreased by more than 53%, the patient was included in the response cohort. If the FAPI-PET/CT results showed that the SUVmax of the primary lesion decreased by less than 53%, remained unchanged or even increased, the patient was placed in the non-response cohort and received concurrent chemoradiotherapy.

SUMMARY:
This study was a single-arm, two-cohort, phase II trial aimed at evaluating the efficacy and safety of FAPI-PET/CT response for guiding the selection of neoadjuvant treatment modes after chemotherapy combined with immunotherapy.

DETAILED DESCRIPTION:
After signing the informed consent form, patients initially underwent two cycles of neoadjuvant chemotherapy in combination with immunotherapy. The chemotherapy protocol consisted of albumin-bound paclitaxel (260mg/m2, with a maximum dose of 400mg) + carboplatin (AUC = 5). Sintilimab was employed for immunotherapy at a fixed dose of 200mg.

FAPI-PET/CT was carried out between days 15 and 22 following two cycles of chemoimmunotherapy. If the FAPI-PET/CT results indicated that the SUVmax of the primary tumor decreased by more than 53%, the patient was included in the response cohort and continued to receive one or two cycles of neoadjuvant chemotherapy combined with immunotherapy after day 22 after the second chemotherapy, every 3 cycles. The chemotherapy and immunotherapy regimens were the same as those in the first and second cycles. After the completion of three to four cycles of chemotherapy combined with immunotherapy, CT was reviewed, and the resectability was evaluated by surgery. For operable patients, surgical resection would be performed within 4 to 6 weeks.

If the FAPI-PET/CT results indicated that the SUVmax of the primary lesion decreased by less than 53%, remained unaltered or even increased, the patient was included in the non-response cohort and received concurrent chemoradiotherapy. At the 4th week of concurrent chemoradiotherapy (18 - 23 fractions of radiotherapy), the resectability was assessed through surgery. For operable patients, surgical resection would be carried out within 4 to 6 weeks after the completion of chemoradiotherapy.

Patients who failed to achieve pCR after surgery will receive adjuvant sintilimab at a dose of 200mg every 3 weeks for one year.

The pCR rate, MPR rate, DFS, OS, FAPI-PET/CT response rate, incidence of postoperative anastomotic leakage, incidence of pneumonia, and quality of life evaluation were observed in patients with or without FAPI response. Meanwhile, the correlation between PD-L1 expression level and PET/CT response was explored, and the feasibility of FAPI-PET/CT response in guiding the selection of neoadjuvant therapy was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Be able to understand and voluntarily provide written informed consent before any procedures required for the study are performed.
* Age between 18 and 75 years.
* Eastern Cooperative Oncology Group (ECOG) performance status score 0-1.
* Histologically confirmed esophageal squamous cell carcinoma.
* T1N1-3M0 or T2-4aNanyM0 as determined by endoscopic ultrasound (EUS) or magnetic resonance imaging (MRI) and PET/CT. All lesions, including tumor and lymph nodes, were required to be resectable.
* Tumors with strong FAPI uptake on baseline PET/CT scan should have a maximum standardized uptake value (SUVmax) ≥5.0.
* Subjects were required to provide preoperative paraffin blocks or white slides of tumor tissue, or freshly collected samples, including at least 3 unstained FFPE pathological slides.
* Female subjects of childbearing potential must have a urine or serum pregnancy test with a negative result within 3 days before the first dose. If urine testing could not confirm the negative result, serum testing was required. Participants who had sex with an unsterilized male partner were required to use an effective contraceptive method from the time of screening and to agree to continue using a contraceptive method for 120 days after the last dose. Discontinuation of contraception after 120 days was discussed with the investigator.
* Unsterilized male subjects who have sex with a female partner of childbearing potential are required to use effective contraception from the time of screening until 120 days after the last dose; Discontinuation of contraception after 120 days is also discussed with the investigator.
* Laboratory tests must meet the following criteria:

Absolute neutrophil count (ANC) ≥ 1500 /µL Platelet count ≥ 100,000/µL Total bilirubin ≤ 2.5 times the upper limit of normal Creatinine clearance (calculated by the following formula) ≥ 60 mL/ minute AST/ALT ≤ 1.5 times the upper limit of normal The modified Cockcroft-Gault equation was used to estimate creatinine clearance (Clcr) : **

For serum creatinine concentration (Sr Cr) expressed in mg/dL:

Clcr (mL/min) = (140-age) × actual weight (kg)/(72 × Sr Cr(mg/dL)) Results for women were calculated using 85% of the Clcr values for men.

Exclusion Criteria:

* A history of malignant tumors within the past five years prior to registration (excluding basal cell carcinoma, squamous cell skin cancer, carcinoma in situ of the bladder, or cervical cancer). Patients who have undergone surgical treatment and have remained disease-free for over five years are still eligible for inclusion.
* Known contraindications include severe allergic reactions to taxanes, platinum-based drugs, 5-FU medications, etc.
* Patients with a documented history of severe allergic reactions to sintilimab.
* Patients who are unwilling or unable to adhere to visit schedules, treatment plans, laboratory tests, and other study requirements.
* Previous radiotherapy administered to the chest or abdomen.
* Patients who have received treatments involving platinum agents, taxanes, 5-FU drugs or PD-1 inhibitors.
* T4 stage tumors exhibiting definite invasion into the spine, heart, major blood vessels or tracheobronchial tree.
* Patients with confirmed cervical or supraclavicular lymph node metastasis or other metastatic lymph nodes that cannot be included in the radiotherapy field nor removed during esophagectomy.
* Patients diagnosed with distant metastases through PET/CT scans or other examinations indicating liver, lung or bone metastases.
* Individuals suffering from significant uncontrolled cardiovascular diseases (such as heart failure), severe coronary artery disease or recent myocardial infarction; also includes those with serious conditions affecting liver or kidney function (e.g., renal insufficiency or liver cirrhosis).
* History of severe central nervous system disorders or mental health issues that may impact treatment compliance and study monitoring.
* Individuals presenting severe surgical contraindications that render them unable to tolerate surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
pCR | up to 12 weeks
  Based on the FAPI-PET/CT responders after chemoradiotherapy, the pCR rate of the continued neoadjuvant chemoradiotherapy was over 44%
pCR | up to 12 weeks
  Patients with a poor FAPI-PET/CT response after chemoradiotherapy were shifted to concurrent chemoradiotherapy, and the pCR rate was no less than 22%.

SECONDARY OUTCOMES:
MPR | up to 12 weeks
  The MPR rate of patients responding to neoadjuvant chemoradiotherapy and FAPI-PET/CT after chemoradiotherapy was based on the MPR rate of patients who continued neoadjuvant chemoradiotherapy, and the MPR rate of patients with a poor FAPI-PET/CT response was converted to concurrent chemoradiotherapy.
DFS | 1 year
  Disease-free survival. Patients responding to neoadjuvant chemoradiotherapy based on FAPI-PET/CT after chemoradiotherapy had a higher 1-year DFS rate than those not responding.
OS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Overall survival
FAPI-PET/CT response rate | At the end of Cycle 2(each cycle is 21 days)
  The proportion of patients with a change in tumor metabolic activity ≥53% (PET/CT response rate) was evaluated by comparing PFAPI-ET/CT results after chemoradiotherapy as an early predictor of response.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Privacy